CLINICAL TRIAL: NCT02557750
Title: Combined Modality Therapy in Hepatoblastoma: South Egypt Cancer Institute Experience
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Morsy, MD, Lecturer, Pediatric Oncology Department, Assiut University
Other Study IDs: Comb Mod Hepatoblastoma SECI
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Hepatoblastoma
Keywords: Childhood Cancer; Pediatric Oncology
MeSH Terms: conditions — Hepatoblastoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to retrospectively investigate the effect of combined modality treatment of pediatric hepatoblastoma and the factors affecting the prognosis in accordance with the experience at the pediatric oncology department at South Egypt Cancer Institute.

DETAILED DESCRIPTION:
Background:

Hepatoblastoma (HB) is the most common malignant liver tumor in children, with an incidence of 0.7 to 1 per million children <15 years of age. Till 1970s, surgery was the primary modality of treatment of HB. Unfortunately, up to 60% of the patients present in an unresectable stage. Later, the chemo- responsiveness of the tumor was demonstrated which led to the incorporation of adjuvant chemotherapy with cisplatinum and doxorubicin in the treatment of HB. International Society of Pediatric Oncology (SIOP) pioneered the concept of neoadjuvant chemotherapy in the management of HB.

Patients & Methods:

In the period from 2002 January till 2016 January, retrieval & analysis of the medical records of pediatric patients with hepatoblastoma will be made at the pediatric oncology department, South Egypt Cancer Institute which represents the largest referral center in Upper Egypt. After pathologic confirmation of the diagnosis, these data will be categorized according to patients' demographics, presenting features, laboratory studies, including tumor markers & histologic subtype, radiographic evaluation, disease staging, treatment course given, and subsequent treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age less than 19 years.
* Patients diagnosed with hepatoblastoma.

Exclusion Criteria:

* Patients whose age more than 18 years.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric cancer patients, those diagnosed with hepatoblastoma, in the period from 2002 January till 2016 January, and received treatment at the pediatric oncology department, their medical records will be retrospectively reviewed for data collection.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2016-01; Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Participants will be retrospectively followed forward in time from the date of initiation of treatment till the primary completion date of the study, an expected average of 5 years
  Time from the date of initiation of treatment until death from any cause
Event Free Survival (EFS) | Participants will be retrospectively followed forward in time from the date of initiation of treatment till the primary completion date of the study, an expected average of 5 years
  Time from the date of initiation of treatment until disease progression, or death for any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Bu, M., D. Terrada, et al. (2006).
- [Background] Douglass EC, Reynolds M, Finegold M, Cantor AB, Glicksman A. Cisplatin, vincristine, and fluorouracil therapy for hepatoblastoma: a Pediatric Oncology Group study. J Clin Oncol. 1993 Jan;11(1):96-9. doi: 10.1200/JCO.1993.11.1.96. PMID 8380296
- [Background] Exelby PR, Filler RM, Grosfeld JL. Liver tumors in children in the particular reference to hepatoblastoma and hepatocellular carcinoma: American Academy of Pediatrics Surgical Section Survey--1974. J Pediatr Surg. 1975 Jun;10(3):329-37. doi: 10.1016/0022-3468(75)90095-0. PMID 49416
- [Background] Mann JR, Kasthuri N, Raafat F, Pincott JR, Parkes SE, Muir KR, Ingram LC, Cameron AH. Malignant hepatic tumours in children: incidence, clinical features and aetiology. Paediatr Perinat Epidemiol. 1990 Jul;4(3):276-89. doi: 10.1111/j.1365-3016.1990.tb00651.x. PMID 2374747
- [Background] Ortega JA, Krailo MD, Haas JE, King DR, Ablin AR, Quinn JJ, Feusner J, Campbell JR, Lloyd DA, Cherlow J, et al. Effective treatment of unresectable or metastatic hepatoblastoma with cisplatin and continuous infusion doxorubicin chemotherapy: a report from the Childrens Cancer Study Group. J Clin Oncol. 1991 Dec;9(12):2167-76. doi: 10.1200/JCO.1991.9.12.2167. PMID 1720452
- [Background] Pritchard J, Brown J, Shafford E, Perilongo G, Brock P, Dicks-Mireaux C, Keeling J, Phillips A, Vos A, Plaschkes J. Cisplatin, doxorubicin, and delayed surgery for childhood hepatoblastoma: a successful approach--results of the first prospective study of the International Society of Pediatric Oncology. J Clin Oncol. 2000 Nov 15;18(22):3819-28. doi: 10.1200/JCO.2000.18.22.3819. PMID 11078495
- [Background] Quinn JJ, Altman AJ, Robinson HT, Cooke RW, Hight DW, Foster JH. Adriamycin and cisplatin for hepatoblastoma. Cancer. 1985 Oct 15;56(8):1926-9. doi: 10.1002/1097-0142(19851015)56:83.0.co;2-g. PMID 2411381
- [Background] von Schweinitz D, Byrd DJ, Hecker H, Weinel P, Bode U, Burger D, Erttmann R, Harms D, Mildenberger H. Efficiency and toxicity of ifosfamide, cisplatin and doxorubicin in the treatment of childhood hepatoblastoma. Study Committee of the Cooperative Paediatric Liver Tumour Study HB89 of the German Society for Paediatric Oncology and Haematology. Eur J Cancer. 1997 Jul;33(8):1243-9. doi: 10.1016/s0959-8049(97)00095-6. PMID 9301450